CLINICAL TRIAL: NCT06875011
Title: Percutaneous Needle Technique is Comparable to Open Z-plasty Surgery for Unilateral Tendon Achilles Lengthening in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1000168
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy; Equinus Foot Deformity in Children With Cerebral Palsy; Gait Analysis in Neurological Disorders
Keywords: cerebral palsy; tendon Achilles; open surgery; z-plasty lengthening; needle lengthening technique
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Open z-TAL: Patients with CP who has undergone unilateral Tendon Achilles Lengthening by open z-plasty (open z-TAL)
- Needle PTAL: Patients with CP who has undergone unilateral Tendon Achilles Lengthening by percutaneous needle technique (needle PTAL)

SUMMARY:
This study aims to compare the outcomes of two surgical techniques for Achilles tendon lengthening in ambulatory children with cerebral palsy (CP): the percutaneous needle technique and the traditional open Z-lengthening technique. The primary objective is to evaluate the effectiveness of these techniques in improving ankle dorsiflexion and gait function one year postoperatively. Secondary objectives include assessing postoperative complications, re-rupture rates, and patient satisfaction. The study is designed as a retrospective, matched-pair cohort study, utilizing data from clinical records, 3D gait analysis (3DGA), and structured telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory children with spastic cerebral palsy (unilateral or bilateral).
* Indication for Achilles tendon lengthening confirmed by 3D gait analysis.
* Underwent unilateral either percutaneous needle technique or open Z-lengthening between 2015 and 2022.
* Availability of preoperative and one-year postoperative 3D gait analysis data.
* Informed consent obtained.

Exclusion Criteria:

* Multilevel surgical interventions.
* Previous foot surgeries that alter foot anatomy.
* Non-compliance with rehabilitation protocols or orthotic use.
* Botulinum toxin-A injections in the triceps surae within six months pre- or post-surgery.
* Incomplete or inadequate 3D gait analysis data.
* Lack of informed consent.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This retrospective, matched-pair cohort study investigates the outcomes of percutaneous needle technique versus open Z-lengthening for Achilles tendon lengthening in children with spastic cerebral palsy. The study will assess changes in ankle dorsiflexion, gait function, and the incidence of postoperative complications. Data will be gathered from 3D gait analysis reports, clinical records, and structured telephone interviews. The primary outcome is the degree of passive ankle dorsiflexion one year postoperatively. Secondary outcomes include active ankle dorsiflexion, adverse events and re-rupture rates. The results aim to inform clinical decision-making and optimize surgical management for children with CP-related gait impairments.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Passive Ankle Dorsiflexion (Degrees) | Measured with the knee extended at one year postoperatively.
  Passive Ankle Dorsiflexion (Degrees) measured with the knee flexed.

SECONDARY OUTCOMES:
Active Ankle Dorsiflexion (Degrees) | Measured with the knee extended at one year postoperatively.
  Active Ankle Dorsiflexion (Degrees): Measured with the knee extended and flexed.
Maximum Ankle Dorsiflexion in Stance Phase | Measured with the knee extended at one year postoperatively.
  Maximum Ankle Dorsiflexion in Stance Phase: Kinematic analysis during 3D gait analysis.
Propulsive Power in Terminal Stance | Measured with the knee extended at one year postoperatively.
  Propulsive Power in Terminal Stance: Measured in watts per kilogram using kinetic analysis.
Postoperative Complications | Measured with the knee extended at one year postoperatively.
  Postoperative Complications: Incidence of infections, hematoma, and re-ruptures within the first postoperative year.

CONTACTS AND LOCATIONS:
Locations (1):
- Vestreviken, Drammen, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: No